CLINICAL TRIAL: NCT06982794
Title: 'UROLIFE': a Patient-Directed Mobile Tool to Streamline the QoL Assessment and Monitoring in Urothelial Carcinoma
Brief Title: A Patient-Directed Mobile Tool to Streamline the QoL Assessment and Monitoring in Urothelial Carcinoma
Acronym: Urolife
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Brigida Anna Maiorano, Principal Investigator, Department of Medical Oncology, IRCCS San Raffaele
Other Study IDs: URO-B01-step1
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma (UC)
Keywords: Quality of life; Self-education; Educational; Urothelial carcinoma; Web-app; Mobile tool; Design-thinking
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with urothelial carcinoma candidate to receive systemic therapy, having a mobile device: Patients will receive a researcher-made questionnaire to gather the demographic and clinical characteristics of the respondents (age, sex, educational level, employment status, type of treatment for UC, physical activity, familiarity and caregiver status, interest, and comfortability with mobile devices and apps).
  Paper questionnaires containing the main contents to be included in the future development of the 'Urolife' web-app will be presented. Four categories of educational and self-management contents will be proposed: 1. Quality of life questionnaires; 2. Self-education on symptoms and AEs tool; 3. Links to verified patients' forums and support organizations for UC; 4. Educational videos and podcasts. Patients will have the opportunity to propose other useful tools. Each tool will be rated by the patients. User needs will be elicited through co-creation sessions held with the Design Thinking method.

SUMMARY:
The goal of this observational study is to select contents and tools for the future development of a web app aiming to support patients' navigation for empowering decision-making through a higher awareness of urothelial carcinoma and its treatments, improving also educational aspects.

The main question it aims to answer is:

What are the contents that patients diagnosed with urothelial carcinoma find useful to include in a web app to streamline their quality of life assessment and monitoring?

Participants candidate for systemic treatments, or already under treatment, will answer questionnaires about the tools to include in a web app designed for urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of urothelial carcinoma;
* ≥ 18 years old,
* candidate for systemic treatment with chemotherapy, immune-checkpoint inhibitors, antibody-drug conjugates, or target therapy (patients can be enrolled also if the treatment has started),
* possession of a mobile device (e.g., smartphone or personal computer) with the physical and psychological ability to use mobile devices,
* understanding and speaking the Italian language,
* ability to sign an informed consent.

Exclusion Criteria:

* not possession of a mobile device,
* unwillingness to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of urothelial carcinoma and candidate to receive systemic treatments at the Ospedale San Raffaele Department of Medical Oncology, Milan (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation score for the Web App contents | 3 months
  A paper questionnaire will be administered to the participants. Each question will regard the description of the tool, with functions and characteristics, to be included in the Web App: 1. Quality of life questionnaires; 2. Self-education on symptoms and adverse events tool; 3. Links to verified patients' forums and support organizations for UC; 4. Educational videos and podcasts. Each section will receive an evaluation of 0 (not interesting), 1 (of moderate interest), or 2 (very interesting). A total score of the questionnaires will determine patients' interest in the different contents. A final free-text section will be given for further patients' purposes not included in the main questionnaire.

SECONDARY OUTCOMES:
eHealth Literacy Scale Score | 3 months
  The eHEALS is an 8-item measure of eHealth literacy developed to measure consumers' combined knowledge, comfort, and perceived skills about the use of mobile device. Each patient will be required to complete the paper questionnaire, and final scores for each questions will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be used only for publication in an aggregate form, and to build a web app. A subsequent phase of the project will be submitted, including the full version of IPD and their sharing agreement.